CLINICAL TRIAL: NCT03073785
Title: A Randomized Phase II Study of the Efficacy and Safety of Hypofractionated Stereotactic Radiotherapy and 5FU or Capecitabine With and Without Zometa in Patients With Locally Advanced Pancreatic Adenocarcinoma
Brief Title: Hypofractionated Stereotactic Body Radiation & Fluorouracil or Capecitabine for Locally Advanced Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0552-16-FB; NCI-2016-01360 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2017-02-28; First posted 2017-03-08 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Adenocarcinoma; Recurrent Pancreatic Carcinoma; Stage I Pancreatic Cancer AJCC v6 and v7; Stage IA Pancreatic Cancer AJCC v6 and v7; Stage IB Pancreatic Cancer AJCC v6 and v7; Stage II Pancreatic Cancer AJCC v6 and v7; Stage IIA Pancreatic Cancer AJCC v6 and v7; Stage IIB Pancreatic Cancer AJCC v6 and v7; Stage III Pancreatic Cancer AJCC v6 and v7; Stage IV Pancreatic Cancer AJCC v6 and v7
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Fluorouracil; dehydroftorafur; Radiosurgery; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (chemotherapy, radiation therapy) (Active Comparator): Participants undergo hypofractionated stereotactic body radiation therapy in 5 fractions on days 1-5. Participants receive fluorouracil IV over 24 hours on day 1 weekly for 4 weeks or capecitabine by mouth every 12 hours starting the evening before day 1 of radiation therapy for 4 weeks as per standard of care. Participants then undergo surgery 6-8 weeks after completion of radiation therapy.
  Interventions: Drug: Capecitabine; Drug: Fluorouracil; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Radiation: Stereotactic Body Radiation Therapy
- Arm B (zoledronic acid, chemotherapy, radiation therapy) (Experimental): Participants receive zoledronic acid IV over a minimum of 15 minutes 1 week prior to radiation therapy. Participants undergo hypofractionated stereotactic body radiation therapy and receive treatment with fluorouracil IV or capecitabine by mouth as in Arm A. Participants then undergo surgery 6-8 weeks after completion of radiation therapy.
  Interventions: Drug: Capecitabine; Drug: Fluorouracil; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Radiation: Stereotactic Body Radiation Therapy; Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Capecitabine — Given by mouth (PO)
  Other Names: Ro 09-1978/000; Xeloda
Drug: Fluorouracil — Given Intravenously (IV)
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Radiation: Stereotactic Body Radiation Therapy — Undergo hypofractionated stereotactic radiotherapy
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
Drug: Zoledronic Acid — Given IV
  Other Names: [1-Hydroxy-2-(1H-imidazol-1-yl)ethylidene]bisphosphonic Acid; CGP 42446; CGP42446A; NDC-Zoledronate; Reclast; ZOL 446; Zometa
  Arms: Arm B (zoledronic acid, chemotherapy, radiation therapy)

SUMMARY:
Pancreatic cancer, most commonly adenocarcinoma, is the fourth leading cause of cancer death in the United States. The mainstay of management centers on surgical resection (if resectable) and although low (15% to 20%), resectability rates are associated with dismal survival. An estimated 80% to 85% of the patients recur after surgical resection, leading to a median survival of 20 to 24 months and potentially even less depending on lymph nodal involvement or positive margins. The rationale for utilizing neoadjuvant therapy, commonly fluoropyrimidine-based or gemcitabine based chemotherapy or Chemoradiotherapy (CRT), involves possibly down staging borderline resectable and unresectable patients, potentially making them resectable candidates.

This randomized phase II trial will study how well hypofractionated stereotactic body radiation therapy (SBRT) and fluorouracil or capecitabine with or without zoledronic acid work in treating participants with pancreatic cancer that has spread to nearby tissue or lymph nodes. Hypofractionated stereotactic body radiation therapy is a specialized radiation therapy that sends higher doses of x-rays over a shorter period of time directly to the tumor using smaller doses over several days which may cause less damage to normal tissue. Drugs used in chemotherapy, such as fluorouracil and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Zoledronic acid is used in cancer patients to reduce cancer symptoms and may make tumor cells more sensitive to radiation. Giving hypofractionated stereotactic body radiation therapy and fluorouracil or capecitabine with or without zoledronic acid may work better in treating pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer, most commonly adenocarcinoma, is the fourth leading cause of cancer death in the United States. The mainstay of management centers on surgical resection (if resectable) and although low (15% to 20%), resectability rates are associated with dismal survival. An estimated 80% to 85% of the patients recur after surgical resection, leading to a median survival of 20 to 24 months and potentially even less depending on lymph nodal involvement or positive margins. The rationale for utilizing neoadjuvant therapy, commonly fluoropyrimidine-based or gemcitabine based chemotherapy or Chemoradiotherapy (CRT), involves possibly down staging borderline resectable and unresectable patients, potentially making them resectable candidates.

This randomized phase II trial will study how well hypofractionated stereotactic body radiation therapy (SBRT) and fluorouracil or capecitabine with or without zoledronic acid work in treating participants with pancreatic cancer that has spread to nearby tissue or lymph nodes. Hypofractionated stereotactic body radiation therapy is a specialized radiation therapy that sends higher doses of x-rays over a shorter period of time directly to the tumor using smaller doses over several days which may cause less damage to normal tissue. Drugs used in chemotherapy, such as fluorouracil and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Zoledronic acid is used in cancer patients to reduce cancer symptoms and may make tumor cells more sensitive to radiation. Giving hypofractionated stereotactic body radiation therapy and fluorouracil or capecitabine with or without zoledronic acid may work better in treating pancreatic cancer.

The primary study objective is to evaluate the efficacy of hypofractionated radiation therapy concurrently with zoledronic acid (Zometa) and fluorouracil or capecitabine. Other study objectives include examining the toxicity of Zometa when used concurrently with hypofractionated radiation therapy, evaluating local failure-free survival and overall survival, determining surgical resection and tumor response rates, measuring Zometa pharmacokinetics, evaluating tumor and organ motion and determining the effect those on the dosimetry, local control and survival. Post-treatment follow-up is for 30 days, then every 3 months for the first year, every 4 months for the second year, and every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed pancreatic adenocarcinoma, either initially diagnosed or recurrent locally advanced disease. The maximum dimension of the treatment target must be =<10 cm. Locally advanced disease defined as: T 1-2N+MO or T3-4 NxMo, or borderline resectable and unresectable adenocarcinoma without distant metastatic disease or resectable T3-4 NxMo disease or M1 with controlled distant disease
* Inoperable conditions with resectable disease (T1-2NoMo)
* Karnofsky performance status of 60% or better. Received recent chemotherapy for pancreatic cancer or completed chemotherapy > 5 years ago for malignancies other than pancreatic cancer with no evidence of the second malignancy at study entry
* Radiation therapy completed > 5 years ago for malignancies other than pancreatic cancer and whose radiation therapy field is not overlapping with the 20% isodose line of current radiation field and no evidence of the second malignancy at study entry
* All malignant disease must be able to be encompassed within a single irradiation field
* Absolute neutrophil count (ANC) greater than or equal to 1500/uL
* Radiographically assessable disease
* Platelet count greater than or equal to 100,000/uL
* Serum creatinine less than or equal to 2.0 mg/dL and total bilirubin less than or equal to 2.0 mg/dL in the absence of biliary obstruction. If biliary obstruction is present, biliary decompression will be required, either endoscopic placement of a biliary stent or percutaneous transhepatic. Once biliary drainage has been established, institution of protocol therapy may proceed when the total bilirubin falls to 4.0 mg/dL or lower
* Calculated creatinine clearance of >= 35.
* Awareness of the neoplastic nature of his/her disease and willingly provide written, informed consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts

Exclusion Criteria:

* Known allergy to Zometa or to anti-emetics appropriate in conjunction with protocol-directed therapy
* Uncontrolled inter-current illness that might jeopardize the ability of the subject to receive the protocol therapy with reasonable safety. This may include, but not limited to, ongoing or active infection requiring intravenous antibiotics, symptomatic congestive heart failure, unstable angina pectoris, or serious, uncontrolled cardiac arrhythmia
* Pregnant and nursing women
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, adequately treated non-invasive carcinomas, or be disease-free for at least 5 years from other cancers
* Active duodenal ulcer or bleeding or history of a gastrointestinal fistula or perforation or other significant bowel problems (severe nausea, vomiting, inflammatory bowel disease and significant bowel resection)
* Known human immunodeficiency virus (HIV) infection, or hepatic insufficiency
* Not currently receiving or have received Zometa within 3 weeks prior to study treatment with Zometa

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Local control With and Without Zometa at Four Months in Follow-up | At 4 months in follow-up
  Local control of tumor will be determined by four dimensional (4D) computed tomography (CT) scans and comparison made between participants receiving Zometa and those who don't.
Local control With and Without Zometa at Eight Months in Follow-up | At 8 months in follow-up
  Local control of tumor will be determined by four dimensional (4D) computed tomography (CT) scans and comparison made between participants receiving Zometa and those who don't.
Local control With and Without Zometa at Twelve Months in Follow-up | At 12 months in follow-up
  Local control of tumor will be determined by four dimensional (4D) computed tomography (CT) scans and comparison made between participants receiving Zometa and those who don't.

SECONDARY OUTCOMES:
Maximum Tolerated Dose of Zoledronic Acid | Up to 30 days after surgery
  Maximum tolerated dose of zoledronic acid will be determined by dose limiting toxicities according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Safety variables to be analyzed are adverse events (AE) and serious adverse events (SAE). AEs and SAEs will be tallied for overall frequency (number and percentage of subjects), worst reported severity, and relationship to study drugs.
Local Failure-free Survival With and Without Zometa | From date of administration of study drug to the date of local failure, assessed up to 5 years
  Time to local failure (disease progression or recurrence determined by imaging, or death) will be analyzed using Kaplan-Meier method between participants receiving Zometa and those who don't.
Overall Survival With and Without Zometa | From date of administration of study drug to the date of death, assessed up to 5 years
  Time to death will be analyzed using Kaplan-Meier method between participants receiving Zometa and those who don't.
Surgically Complete Resection Rate With and Without Zometa | Immediately after surgery
  The number and proportion of participants undergoing complete resection (negative margin) will be determined between participants receiving Zometa and those who don't.
Pathologic Response After Resection With and Without Zometa | Immediately after surgery
  The pathologic response will be scored from 0-9 by a pathologist, 0 is no response and 9 is complete response between participants receiving Zometa and those who don't.
Change in Tumor Size after Stereotactic Body Radiation Therapy With and Without Zometa | Within 1 month prior to SBRT and 4-5 weeks after SBRT
  Tumor size will be measured on computed tomography (CT)/magnetic resonance imaging (MRI) before and after stereotactic body radiation therapy (SBRT) and compared between participants receiving Zometa and those who don't.
Change of maximum and average Standardized Uptake Values after Stereotactic Body Radiation Therapy With and Without Zometa | Within 1 month prior to SBRT and 4-5 weeks after SBRT
  The maximum and average standardized uptake values SUV will be measured on Positron Emission Tomography (PET) before and after Stereotactic Body Radiation Therapy (SBRT) and will be compared between participants receiving Zometa and those who don't.
Tumor and Organ Motion | Immediately prior to stereotactic body radiation therapy (SBRT)
  The amplitude of 3D tumor/organ motion will be measured using four dimensional (4D) computed tomography (CT) scans.

OTHER OUTCOMES:
RNA Sequence Assessment of Gene Expression of Cholesterol Biosynthesis for Resection With or Without Zometa | Up to 5 years
  Change in expression of genes involved in cholesterol biosynthesis in participants who undergo resection will be assessed between participants receiving Zometa and those who don't.
Pharmacokinetics of Zoledronic Acid | At 0 and 1 hours post-zoledronic acid dose, and before stereotactic body radiation therapy (SBRT) treatments on days 2, 3, 4, and 5
  The concentration of plasma zoledronic acid will be measured in participants who received zoledronic acid.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Lin, MD, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No